CLINICAL TRIAL: NCT00748059
Title: The Pathophysiology of Orthostatic Hypotension
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Emily M. Garland, Research Associate Professor, Vanderbilt University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 030752; HL056693
Record Dates: First submitted 2008-09-05; First posted 2008-09-08 (Estimated); Last update posted 2021-05-12 (Actual); Status verified 2021-05

CONDITIONS: Autonomic Nervous System Diseases; Orthostatic Hypotension; Dopamine Beta-Hydroxylase Deficiency; Orthostatic Intolerance
Keywords: autonomic nervous system diseases; blood pressure; congenital; orthostasis; catecholamines
MeSH Terms: conditions — Autonomic Nervous System Diseases; Hypotension, Orthostatic; dopamine beta hydroxylase deficiency; Orthostatic Intolerance; Dizziness | interventions — Standing Position; Phenylephrine; Clonidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): Patients with Orthostatic Hypotension
  Interventions: Procedure: Standing or upright tilt; Procedure: Microneurography; Procedure: QSweat; Device: neck cuff stimulation; Drug: phenylephrine,isoproterenol,nitroprusside,propranolol,edrophonium,atropine,tyramine; Drug: clonidine,yohimbine,metoclopramide,alpha-methyldopa; Procedure: BodPod; Procedure: Eye exam; Procedure: Sleep study; Procedure: Pain response testing; Procedure: Metabolic chamber; Procedure: Brain function studies; Procedure: Bicycle Exercise Test

INTERVENTIONS:
Procedure: Standing or upright tilt — stand upright or tilt table test
Procedure: Microneurography — Recording from sympathetic nerve
Procedure: QSweat — quantitative sweat testing
Device: neck cuff stimulation — Blood pressure receptors in the neck arteries may be stimulated by applying suction through a collar around the neck.
Drug: phenylephrine,isoproterenol,nitroprusside,propranolol,edrophonium,atropine,tyramine — IV Pharmacological Testing
  phenylephrine 12.5 - 400 ug, isoproterenol 0.1 - 0.4 ug or higher until desired effect, nitroprusside 0.1 - 1.6 ug/kg, propranolol 1.1 mg/min, edrophonium maximum of 10 mg, atropine .01 mg/kg, tyramine 250-4000 ug or higher until desired effect
Drug: clonidine,yohimbine,metoclopramide,alpha-methyldopa — Oral Pharmacological Testing
  clonidine 0.1-0.3 mg, yohimbine 5-10 mg, metoclopramide 10 mg, alpha-methyldopa 62.5 mg, placebo
Procedure: BodPod — Determination of body composition
Procedure: Eye exam — Examination of pressure in the eye and eyelid fatiguability. The following eyedrops might be used:
  1. 0.5% proparacaine (Alcaine, Allergan, Inc)
  2. Fluress (0.4% benoxinate hydrochloride, fluorescein sodium, Akorn, Inc)
  3. 0.5%, 1% tropicamide (Mydriacyl, Alcon)
  4. Over-the-counter preservative-free artificial tears
  5. 0.25%, 2.5% and 10% phenylephrine (Bausch and Lomb)
  6. 1% cyclopentolate hydrochloride (Alcon)
Procedure: Sleep study — Recording of sleep pattern overnight
Procedure: Pain response testing — Subjects will rate the quality and intensity of 2 pain tasks.
Procedure: Metabolic chamber — Determination of metabolic rate via 24hr stay in whole-room indirect calorimeter
Procedure: Brain function studies — Questionnaires and computer tasks, an EEG and an MRI may be used to assess brain function.
Procedure: Bicycle Exercise Test — Blood pressure and heart rate may be monitored while exercising on a stationary bicycle.

SUMMARY:
The purpose of this study is to determine the cause of low blood pressure in selective patients who have problems with their involuntary (autonomic) nervous system. These patients frequently have had symptoms throughout their life, and their disorder might have a genetic basis. The biochemical, physiological and pharmacological procedures in this study should help us define the problem and perhaps lead to more effective treatment.

ELIGIBILITY:
Inclusion Criteria:

* severe orthostatic hypotension and other autonomic symptoms but do not meet criteria for standard diagnosis
* non-smokers
* drug-free
* able to give informed consent
* free of pulmonary, renal, hematopoietic, hepatic and cardiac disease

Exclusion Criteria:

* medications affecting the autonomic nervous system
* any chronic illness
* anemia (Hct<30)
* women of childbearing age who are pregnant or nursing
* smokers

Ages: 12 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 1996-12; Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
hemodynamic changes with standing | following test

SECONDARY OUTCOMES:
blood and urine hormones | after test
blood volume | during supine and/or upright postures
sympathetic nerve activity | during stimulation of sympathetic nervous system
quantitative sweat testing | 2 hours
Eye function | once
Sleep efficiency | once
Metabolic rate | once
Pain response | once
Responses on questionnaires and computer tasks designed to assess brain function | once

CONTACTS AND LOCATIONS:
Overall Officials: Emily M Garland, PhD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States

REFERENCES:
- [Derived] Arnold AC, Garland EM, Celedonio JE, Raj SR, Abumrad NN, Biaggioni I, Robertson D, Luther JM, Shibao CA. Hyperinsulinemia and Insulin Resistance in Dopamine beta-Hydroxylase Deficiency. J Clin Endocrinol Metab. 2017 Jan 1;102(1):10-14. doi: 10.1210/jc.2016-3274. PMID 27778639